CLINICAL TRIAL: NCT03719833
Title: Sentinel Lymph Node Biopsy After Neoadjuvant Oncological Treatment in Luminal B, HER-2 Positive and Triple Negative Breast Cancer Patients in Stage T1-3 N0-2 M0 at the Time of Diagnose
Brief Title: Sentinel Lymph Node Biopsy After Neoadjuvant Treatment in Breast Cancer Patents
Status: Completed | Type: Observational
Sponsor: Clinical Hospital Center Rijeka (Other)
Responsible Party: Principal Investigator, Ana Car Peterko, general surgeon, surgical oncologist, FEBS, CEBS, Clinical Hospital Center Rijeka
Other Study IDs: SLNB-ACP
Record Dates: First submitted 2018-10-23; First posted 2018-10-25 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Sentinel Lymph Node Biopsy; Neoadjuvant Chemotherapy
Keywords: Breast Cancer; Sentinel Lymph Node Biopsy; Neoadjuvant Chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (3):
- 1-control group-T1-T2 N0 M0: Breast cancer patients in T1 N0 M0 stage at the time of diagnosis who initially undergo surgical treatment (quadrantectomy/mastectomy + sentinel lymph node biopsy).
  All patients will be followed for 5 years after surgery
- 2-T2-T3 N0 M0: Breast cancer patients in the T2-T3 N0 M0 stage at the time of diagnosis who undergo neoadjuvant oncological treatment followed by surgery (quadrantectomy/mastectomy + sentinel lymph node biopsy). For the presence of any residual tumour in lymph node(s) at the final pathology report, ALND will be performed.
  All patients will be followed for 5 years after surgery
- 3-T1-T3 N1-N2 M0: Breast cancer patients in T1-T3 N1-N2 M0 stage at the time of diagnosis who undergo neoadjuvant oncological treatment followed by ultrasound reevaluation of axillary lymph nodes that indicate complete clinical axillary remission. The surgical procedure that would be performed is quadrantectomy/mastectomy + sentinel lymph node biopsy.
  Before initiating neoadjuvant treatment biopsy (FNA) proven positive node will be marked with a titanium clip and at the time of surgery removed and pathologically examined regardless presenting as a sentinel node or not.
  For the presence of any residual tumour in lymph node(s) at the final pathology report, ALND will be performed All patients will be followed for 5 years after surgery

SUMMARY:
This clinical trial is designed as an observational study of 8-9 years of overall duration, but the first results and conclusions could be achieved in 3-4 years. In the first phase, which would last 3-4 years, the investigators will form three predetermined groups of breast cancer patients that would be monitored in the second phase for 5 postoperative years.

All patients involved in this trial would undergo a defined protocol. All patients participating in this trial and all members of the investigation team would be completely introduced to the plan and aims of this trial.

Two main hypotheses of this trial are that SLNB does not have a negative impact on clinical outcomes (locoregional recurrence and overall survival) in initially node-positive patients who achieved complete clinically axillary remission after neoadjuvant systemic treatment and that lymph node status after neoadjuvant treatment is a significantly more relevant prognostic factor than nodal status at the time of diagnosis.

Therefore, the aim is to establish that sentinel lymph node biopsy, in node-positive breast cancer patients that achieve clinical remission after neoadjuvant treatment, is a reliable approach for surgical axillary management.

Data would be collected individually for each patient and recorded on appropriate forms. After data completion, the principal investigator would import encoded data into the register. Data collected in this trial would be used for publications.

DETAILED DESCRIPTION:
This clinical trial is designed as a prospective, observational, non-randomized clinical trial of 8-9 years of overall duration, but the first results and conclusions (secondary outcomes) could be achieved in 3-4 years from the beginning of the study.

Based on ultrasound and/or magnetic resonance assessment of primary tumour dimensions, pathological report of core needle biopsy, ultrasound evaluation of axillary lymph nodes and cytologically proven positive lymph nodes, patients would be divided into three predefined groups and would undergo predetermined group protocol.

Group 1 (T1-2 N0 M0) protocol: Surgery is primary treatment (quadrantectomy/mastectomy and sentinel lymph node biopsy).

Group 2 (T2-3 N0 M0) protocol: Neoadjuvant oncological treatment is primary therapy followed by surgery (quadrantectomy/mastectomy and sentinel lymph node biopsy) and afterwards by adjuvant oncological treatment. Before neoadjuvant treatment, all patients would undergo magnetic resonance (MR) imaging and ultrasound-guided placement titanium clip in the primary tumour site. Clinical assessment of the effectiveness of neoadjuvant treatment would be evaluated by breast MR imaging in the middle and at the end of the neoadjuvant systemic treatment.

Group 3 (T1-3 N1-2 M0) protocol includes the Group 2 protocol in addition to FNA (cytology) proof of positive node, ultrasound-guided marking positive node with titanium clip before starting neoadjuvant protocol, ultrasound and MR imaging reevaluation of axillary nodes at the end of neoadjuvant treatment and for those patients who achieve complete clinical remission of axillary lymph nodes, biopsy of marked node would be performed in context of standard surgical procedure (in addition to quadrantectomy/mastectomy and sentinel lymph node biopsy) regardless being sentinel node or not.

For the presence of any size residual tumour in lymph node(s) in groups 2 and 3 axillary lymph node dissection will be performed.

All patients would be controlled periodically in the postoperative five-year follow-up period to determine the prevalence of locoregional recurrence, progression of disease to the M1 stage and overall survival rate.

The results would be compared among groups, to available literature data and our former (historical) data of patients of the same stage but treated in the period from 2011 to 2014 (i.e. without neoadjuvant therapy).

In the first phase, which would last 3-4 years, the investigators would form three predetermined groups of breast cancer patients that would be monitored in the second phase for 5 postoperative years and analyse secondary outcome measures.

According to statistical analysis made of former data of Clinical Hospital Centar Rijeka, groups should be made of at least 30 patients in each group.

All patients participating in this trial and all members of the investigation team would be completely introduced to the plan and aims of this trial.

Two main hypotheses of this trial are that SLNB does not have a negative impact on clinical outcomes (locoregional recurrence and overall survival) in initially node-positive patients who achieved complete clinically axillary remission after neoadjuvant systemic treatment and that lymph node status after neoadjuvant treatment is a significantly more relevant prognostic factor than nodal status at the time of diagnosis.

Therefore, the aim is to establish that sentinel lymph node biopsy, in node-positive breast cancer patients that achieve clinical remission after neoadjuvant treatment, is a reliable approach for surgical axillary management and that does not have a negative impact on the oncological principles and clinical outcomes.

Data would be collected individually for each patient during the diagnostic and therapeutic period and in the follow-up period (periodic ambulance controls) for 5 postoperative years.

Data would be recorded on appropriate forms. After data completion, the principal investigator would import encoded data into the register. All data would be available to all members of the investigation team, members of Ethic Committee and a person in charge of statistic analysis. Data collected in this trial would be used for publications and self-control of our multidisciplinary team for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be female
* Patients must be older than 18 years of age and younger than 80 years of age
* Patients must have biopsy-proven breast cancer, histological type-ductal, immunophenotype-Luminal B, HER-2 positive and triple-negative
* Patients with nodal disease (N1-N2) must have fine needle aspiration proven positive node and marked node with titanium clip before onset of neoadjuvant treatment
* Patients treated (oncological and surgical) in Clinical Hospital Centar Rijeka from September 2018 till May 2022
* Patients must be in stage cT1-3 cN0-2 cM0 at the time of diagnosis and cN0 at the time of the surgery
* Patients that are eligible for neoadjuvant oncological treatment, accepting to undergo it and complete it
* Patients who understand, accept and have signed the approved consent form

Exclusion Criteria:

* Patents in T4 stage and/or N3 stage and/or M1 stage at the time of diagnosis
* Patients with inflammatory carcinoma
* Patients with bilateral disease
* Patients with ipsilateral recurrence
* Patients with histological type-lobular and immunophenotype-Luminal A
* Patients that are not eligible for oncological treatment according to protocol, either neoadjuvant or adjuvant, or oncological treatment was interrupted (aborted or completed in another institution)
* Patients that have had previously SLNB or ALND or radiotherapy to the axillary nodes
* Patients that have been or are treated for other malignant disease
* Patients with hypersensitivity or allergy to radiocolloid
* Patients without complete documentation required for this study
* Pregnant patients
* Psychiatric patients
* Male patients

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Groups will be formed of the breast cancer patients who meet the eligible criteria treated in Clinical Hospital Centar Rijeka in a defined period
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Impact of sentinel lymph node biopsy procedure on locoregional recurrence for group 3 sentinel node negative patients | 5 postoperative years
  Locoregional recurrence for group 3 sentinel node negative patients compared to group 1 and 2, to our former (hystorical) data and literature data
Correlation of sentinel node negative patients from group 3 patients and overall survival | 5 postoperative years
  Overall survival from sentinel node negative patients from group 3 compared to overall survival from sentinel node positive patients from group 3 and overall survival from patients from group 3 that did not achieve complete clinical axillary remission.
  Overall survival for group 3 sentinel node negative patients compared to group 1 and 2 and to our former data (patients of same stage at diagnosis treated without neoadjuvant systemic therapy)
Correlation of sentinel node negative patients from group 3 and disease progression free survival | 5 postoperative years
  Disease progression free survival from sentinel node negative patients from group 3 compared to disease progression free survival from sentinel node positive patients from group 3 and disease progression free survival from patients from group 3 that did not achieve complete clinical axillary remission.
  Disease progression free survival for group 3 sentinel node negative patients compared to group 1 and 2 and to our former data (patients of same stage at diagnosis treated without neoadjuvant systemic therapy)

SECONDARY OUTCOMES:
Evaluate the correlations of axillary response to neoadjuvant treatment and pathological characteristic of tumor | 4 years
  Statistical analysis of treated patients and outcomes of neoadjuvant treatment-analysis of complete pathological axillary remission related to characteristics of primary tumor (type, grade, size, proliferation index and presence of lymphovascular invasion) Evaluate when is nodal disease indication for neoadjuvant treatment regardless the tumor size
Evaluate accuracy of standard breast MR imaging in axillary lymph node evaluation after neoadjuvant treatment (overall and related to tumor subtypes) | 4 years
  Sensitivity, Specificity, Positive Predictive Value and Negative Predictive Value of breast MR imaging in evaluation of axillary lymph nodes after neoadjuvant treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ana Car Peterko, Principal Investigator — Clinical Hospital Centar Rijeka
Locations (1):
- Ana Car Peterko, Rijeka, Croatia, Croatia

IPD SHARING:
Plan to Share IPD: No